CLINICAL TRIAL: NCT04391595
Title: A Phase 0/2 Study of LY3214996 (ERK Inhibitor) in Combination With Abemaciclib (CDK4 and 6 Inhibitor) in Recurrent Glioblastoma Participants Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration
Brief Title: LY3214996 Plus Abemaciclib in Recurrent Glioblastoma Patients
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Nader Sanai, Deputy Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-07
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma; GBM; Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — abemaciclib; LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): 400 mg of LY3214996 QD for 6 doses and 100 mg of Abemaciclib BID for 11 doses over 5.5 days prior to surgical resection. On Day 6, participants will receive Abemaciclib + LY3214996 dose 7 to 9 hours prior to craniotomy for tumor resection.
  Interventions: Drug: Abemaciclib; Drug: LY3214996

INTERVENTIONS:
Drug: Abemaciclib — 100 mg of Abemaciclib BID for 11 doses over 5.5 days prior to surgical resection. Participants with tumors demonstrating PK-response in Phase 0 will continue treatment with recommended Phase 2 dose (RP2D) continuously in 21d cycles after surgery.
Drug: LY3214996 — 400 mg of LY3214996 daily for 6 doses over 5.5 days prior to surgical resection. Participants with tumors demonstrating PK-response in Phase 0 will continue treatment with recommended Phase 2 dose (RP2D) continuously in 21d cycles after surgery.

SUMMARY:
This trial is an open-label, multicenter, Phase 0/2 trial that will enroll up to 50 participants with recurrent glioblastoma which are schedule for resection. In the lead-in cohort, a total of 10 participants will be enrolled into the proposed phase 0 clinical trial. Participants will be administered LY3214996 plus Abemaciclib prior to surgical resection of their tumor. If positive PK results are demonstrated in ≥50% of Phase 0 participants and at least 5 participants are enrolled into Phase 2, up to approximately 40 additional participants will be enrolled in the dose expansion cohort in order to achieve a total of 25 participants enrolled into Phase 2 (lead-in cohort + dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Prior resection of histologically diagnosed WHO Grade IV glioma defined as glioma participants who have progressed on or following standard (Stupp regimen) therapy, which included maximal surgical resection, temozolomide, and fractionated radiotherapy.
2. Recurrence must be confirmed by diagnostic biopsy with local pathology review or contrast-enhanced MRI.
3. Participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm, as per RANO criteria.
4. Sufficient archival tissue available to confirm eligibility.
5. For gliomas, archival tissue must demonstrate: (a) RB positivity (≥20%) on immunohistochemistry (IHC); or, no RB mutations on next-generation sequencing (NGS), (b) Chromosomal loss of CDKN2A/B/C; or, CDK4/6 amplification on array CGH or NGS, (c) pERK positivity (>30%) on IHC.
6. Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
7. Participant has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative(s), and assent if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
9. Age ≥18 at time of consent
10. Have a performance status (PS) ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale (Oken et al. 1982)
11. Ability to swallow oral medications.
12. Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

    Adequate bone marrow function:
    * absolute neutrophil count ≥1,000/mcL
    * platelets (at time of surgery) ≥100,000/mcL
    * hemoglobin ≥8.0 g/dL Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.

    Adequate hepatic function:
    * total bilirubin ≤1.5 X ULN Participants with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
    * AST(SGOT) ≤3 X institutional ULN
    * ALT(SGPT) ≤3 X institutional ULN
13. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
14. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 months after the end of treatment administration.
15. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and for an additional 6 months after the end of treatment administration.
16. Agreement to adhere to Lifestyle Considerations throughout study duration
17. Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Day 1. A washout period of at least 21 days is required between last chemotherapy dose and Day 1 (provided the patient did not receive radiotherapy).
18. Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and Day 1.

Exclusion Criteria:

1. Current use of coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
2. Pregnancy or lactation.
3. Known allergic reactions to components of the abemaciclib or LY3214996.
4. Active infection or fever >38.5°C requiring systemic antibiotic, antifungal or antiviral therapy within 4 weeks of Day 1.
5. Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis.
6. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
7. Have history of central or branch retinal artery or venous occlusion with significant vision loss or other retinal diseases that cause current visual impairment or would likely cause visual impairment over the time period of the study.
8. Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
9. Prior therapy with any CDK4/6 inhibitor or any ERK1/2 inhibitor. Prior therapy is defined as a therapeutic dosing.
10. Treatment with another investigational drug or other intervention within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
11. Have a mean QT interval corrected for heart rate (QTc) of ≥470 milliseconds on screening electrocardiogram (ECG) as calculated using the Bazett's formula.
12. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-11 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2028-02-13 (Estimated)

PRIMARY OUTCOMES:
Phase 0: Pharmacokinetic analysis of tumor tissue | 8 hour
  Total and Unbound LY3214996 and Abemaciclib (and related M2 and M20 metabolites) concentration in enhancing and non-enhancing tumor tissue
Phase 0: Pharmacokinetic analysis of cerebrospinal fluid (CSF) | 8 hour
  Total and Unbound LY3214996 and Abemaciclib (and related M2 and M20 metabolites) concentration in CSF
Pharmacokinetic analysis of plasma | Day 6 at 0, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose
  Total and Unbound LY3214996 and Abemaciclib (and related M2 and M20 metabolites) concentration in plasma
Phase 2: Progression-free survival | up to 60 months
  Phase 2: 6-month progression-free survival (PFS6) rate measured from time of surgery to date of recurrence

SECONDARY OUTCOMES:
Phase 0: PD Analysis | Intraoperatively
  Phase 0: percentage of pRSK+, pERK+, pRB+, pFOXM1, MIB-1+ and Cleaved Caspase 3+ cells from the surgical tissue will be quantified and compared to baseline archival tissue.
Number of Adverse Events | up to 30 days after the last study dose
  Number of Adverse Events
Incidence of drug-related toxicity | up to 30 days after the last study dose
  Drug-related toxicity
Incidence of treatment-emergent adverse events | up to 30 days after the last study dose
  Treatment-emergent adverse events
Deaths | up to 60 months
  Deaths
Incidence of clinical laboratory abnormalities per CTCAE | up to 30 days after the last study dose
  Clinical laboratory abnormalities per CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Deputy Director of the Ivy Brain Tumor Center
Locations (3):
- United States (3):
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ivy Brain Tumor Center Website — https://www.ivybraintumorcenter.org/